CLINICAL TRIAL: NCT06005194
Title: Telehealth Delivered Exercise Promotion to Treat Major Depression After TBI: A Randomized Controlled Trial (InMotion)
Brief Title: InMotion - Telehealth Delivered Exercise Promotion to Treat Major Depression After TBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charles Bombardier, Professor of Rehabilitation Medicine, University of Washington, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00017569; 90DPTB0024 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2023-05-18; First posted 2023-08-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: TBI (Traumatic Brain Injury); Depressive Disorder, Major; Clinical Depression; Mood Depressed; Physical Inactivity
Keywords: Exercise Intervention; Traumatic Brain Injury (TBI); Motivational Interviewing; Telehealth
MeSH Terms: conditions — Brain Injuries, Traumatic; Depressive Disorder, Major; Consciousness Disorders; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait List Control (WLC) Condition (Placebo Comparator): The WLC control condition entails following usual care and includes the ability to participate in the intervention at the 12 week-end point for the intervention group. The WLC condition is based on equity considerations; the investigators want all participants to have access to treatment. Equity is especially important given our plans to over-enroll African American persons given statistically increased barriers to access care.
  Interventions: Behavioral: InMotion
- InMotion Intervention Condition (Active Comparator): The intervention consists of a manualized physical activity counseling program and includes motivational interviewing over a HIPAA-compliant telehealth delivery model. There will be 8 counseling sessions over 12 weeks. Sessions will be 30-90 minutes long and scheduled during weeks 1-4, 6, 8, 10, and 12. The Fitbit Charge 5 will be set up to sync with the participants' internet-connected device to share activity data with the physical activity coach /interventionist to monitor progress and tailor treatment goals.
  Given the InMotion intervention was designed to treat Major Depressive Disorder (MDD) in Traumatic Brain Injury (TBI), the intervention will be delivered by a mental health provider (licensed masters level social worker/MSW) with training and supervision in behavioral aspects of exercise promotion and supervised by a psychologist (who is also the study Principal Investigator) and a physical therapist.
  Interventions: Behavioral: InMotion

INTERVENTIONS:
Behavioral: InMotion — A manualized physical activity counseling program that is based on the Diabetes Prevention Program (DPP) that has been adapted for TBI

SUMMARY:
The purpose of this randomized controlled trial is to evaluate whether the InMotion intervention, delivered via telehealth (using a HIPAA-compliant video platform or phone), which uses evidence-based behavioral and motivational counseling to increase daily physical activity, is an effective treatment for Major Depressive Disorder (MDD) for people who are at least one year out from sustaining a traumatic brain injury (TBI). The first aim is to compare the efficacy of the InMotion intervention to the waitlist control (WLC) condition on measures of depression severity and associated conditions in under-active adults with TBI and MDD. For the second aim the investigators plan to identify possible moderators of exercise treatment effects. The third aim will examine possible mediators of treatment outcome. In addition, the weekly dose of exercise, the extent to which exercise generates positive affect, and engagement in enjoyable or meaningful aspects of life will be explored.

DETAILED DESCRIPTION:
Telehealth delivered exercise promotion to treat major depression after traumatic brain injury (TBI): A randomized controlled trial, or InMotion, is a fully-powered, single-blind, randomized controlled trial versus wait-list control (WLC) condition focused on the comparing the InMotion intervention. The intervention is delivered via telehealth and uses evidence-based behavioral and motivational counseling to increase daily physical activity, and is being tested to see whether this can be an effective treatment for Major Depressive Disorder (MDD) for people who are at least one year out from sustaining a traumatic brain injury (TBI). The goal of the study is for all participants to achieve 150 minutes per week of moderate to vigorous physical activity (MVPA), a dose of physical activity already shown to be effective to treat MDD in a healthy population.

The InMotion intervention is a home- and community-based physical activity counseling program based on the widely replicated Diabetes Prevention Program (DPP). The physical activity coach/Interventionist is a mental health provider (Master of Social Work/MSW) who has training and supervision in behavioral aspects of exercise promotion and will use motivational interviewing, telehealth technology using a HIPAA-compliant telehealth delivery model. The intervention also includes the use of a wearable activity monitor (Fitbit activity tracker watch - Charge 5) to facilitate goal setting.

Enrollment into the Traumatic Brain Injury Model System (TBIMS) study is required for eligibility for InMotion. Additionally, this study will capitalize on the infrastructure of the TBIMS for its screening and some data collection.

Specific Aims Aim 1: To compare the efficacy of the InMotion intervention to the waitlist control (WLC) condition on measures of depression severity and associated conditions in under-active adults with traumatic brain injury (TBI) and Major Depressive Disorder (MDD).

Hypothesis 1a: There will be a significantly greater reduction in depression severity as measured by the Symptom Checklist-20 (SCL-20) over 12 weeks in the InMotion intervention group vs. the wait-list control (WLC) group.

Hypothesis 1b: Compared to the WLC group, the InMotion intervention group will demonstrate significantly greater improvement on secondary outcome measures: MDD diagnosis (yes/no), depression remission (yes/no), anxiety, pain, fatigue, and quality of life from baseline to 12-weeks.

Hypothesis 1c: Within the InMotion intervention group, the investigators will describe how much/if any improvement on outcomes is maintained from the end of the treatment period (12 weeks) to follow-up (24 weeks).

Rationale for Aim 1: A statistically significant reduction in depression symptom severity is the most common metric for depression treatment efficacy and what will be used to power the study. However, the investigators also want to assess clinically meaningful changes in depression such as depression diagnosis and depression remission. The investigators will study the impact of the intervention on anxiety, pain, fatigue, and quality of life in people with TBI because these are correlated with depression and important outcomes.

Aim 2: To identify possible moderators of exercise treatment effects. Hypothesis 2: Self-identified race (African American vs. not African American), sex (female vs. male), TBI severity (moderate vs. severe), or concurrent exposure to antidepressant or psychotherapy vs. neither will moderate the effect of InMotion intervention on depression severity.

Rationale for Aim 2: Some participant groups may benefit differentially from exercise.

Identifying factors associated with response to treatment will guide future research.

Aim 3: To identify possible mediators of treatment outcome. Investigators will explore weekly dose of exercise, the extent to which exercise generates positive affect, and engagement in enjoyable or meaningful aspects of life.

Hypothesis 3: The InMotion intervention will be indirectly associated with improved outcomes by its association with higher self-reported weekly minutes/week of activity, higher positive affect, and greater involvement in meaningful activities.

Rationale for Aim 3: Analysis of potential mediators of treatment effects can help guide the refinement of the InMotion intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the Traumatic Brain Injury Model System (TBIMS) from one of the six referring centers.
* Must be between 18-64 years of age at the time of enrollment.
* Must have cognitive capacity to consent.
* Must be >1 year out from the date of the Traumatic Brain Injury.
* Meet the -5 criteria for major depressive disorder (as determined by the Mini International Neuropsychiatric Interview (MINI)).
* Must receive a Health Contribution Score (HCS) of <24 on the Godin Leisure Time Exercise Questionnaire.
* Deemed medically safe to exercise (based on the Physical Activity Readiness Questionnaire (PAR-Q+) modified (if a yes response to any question, physician attestation required).
* Must have a permanent residence and have access to the internet.
* We will over-enroll people who identify as African American because they are at higher risk of depression and face disproportionate barriers to treatment relative to whites. We chose to over-sample African Americans rather other racial or ethnic groups because they represent the second largest racialized subgroup within the full Traumatic Brain Injury Model Systems (18%) and 27% of those with Major Depressive Disorder (MDD). Therefore, we will enroll a sample that is 27% people who identify as African American.

Exclusion Criteria:

* We will exclude people with active suicidal intent or plan or other severe psychiatric conditions (bipolar disorder, schizophrenia, psychosis, any schizoaffective disorder).
* We will exclude people with current substance use disorder (excluding tobacco) because they require intensive treatment, specifically people who report having > 5 drinks for men or >4 for women on a single occasion AND have >14 drinks for males / > 7 drinks per week for females per week. These questions are an existing part of the Traumatic Brain Injury Model System, Form II follow-up interview and participant exclusion for this will take place as part of that study.
* We will exclude people for drug dependence as defined within the Mini International Neuropsychiatric Interview (MINI).
* We will exclude people not fluent in English.
* People with pending surgery or on an unstable dose of standard depression treatment will be deferred until they are recovered or on stable treatment regimens for at least 3 weeks.
* To ensure safety in the trial we will exclude people who have suicide intent or plan and immediately refer them for treatment. We will measure suicide risk at every outcome assessment point and address elevated risk via established assessment and intervention protocols.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Hopkins Symptom Checklist-20 (SCL-20) | Baseline
  The HSCL-20 is a 20-item self-report depression scale on which respondents rate depression symptom severity over the past week on a 5-point scale ranging from (0) not at all to (4) extremely. The total score represents the mean of the 20 items. The total score can range from 0 to 4 with higher numbers indicating worse symptoms.
Hopkins Symptom Checklist-20 (SCL-20) | 12 weeks
  The HSCL-20 is a 20-item self-report depression scale on which respondents rate depression symptom severity over the past week on a 5-point scale ranging from (0) not at all to (4) extremely. The total score represents the mean of the 20 items. The total score can range from 0 to 4 with higher numbers indicating worse symptoms. We will be measuring depression severity at 12 weeks controlling for depression severity at baseline.
Hopkins Symptom Checklist-20 (SCL-20) | 24 weeks
  The HSCL-20 is a 20-item self-report depression scale on which respondents rate depression symptom severity over the past week on a 5-point scale ranging from (0) not at all to (4) extremely. The total score represents the mean of the 20 items. The total score can range from 0 to 4 with higher numbers indicating worse symptoms. We will be measuring depression severity at 24 weeks controlling for depression severity at baseline.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  The PHQ-9 is a 9 item measure of depression severity with excellent sensitivity, specificity and responsiveness in people with TBI and will be used for pre-screening as well as each data collection to calculate minimal clinically important differences (MCID). Each item is rated on a 0 (not at all) to 3 (nearly every day) scale. The total score ranges from 0-27. A higher score indicates increased depression severity.
Patient Health Questionnaire-9 (PHQ-9) | 12 weeks
  The PHQ-9 is a 9 item measure of depression severity with excellent sensitivity, specificity and responsiveness in people with TBI and will be used for pre-screening as well as each data collection to calculate minimal clinically important differences (MCID). Each item is rated on a 0 (not at all) to 3 (nearly every day) scale. The total score ranges from 0-27. A higher score indicates increased depression severity.
Patient Health Questionnaire-9 (PHQ-9) | 24 weeks
  The PHQ-9 is a 9 item measure of depression severity with excellent sensitivity, specificity and responsiveness in people with TBI and will be used for pre-screening as well as each data collection to calculate minimal clinically important differences (MCID). Each item is rated on a 0 (not at all) to 3 (nearly every day) scale. The total score ranges from 0-27. A higher score indicates increased depression severity.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Baseline
  The GLETQ measures number of bouts per week (0-7) of mild, moderate, or strenuous exercise that last at least 15 minutes.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | 12 weeks
  The GLETQ measures number of bouts per week (0-7) of mild, moderate, or strenuous exercise that last at least 15 minutes.
Godin Leisure-Time Exercise | 24 weeks
  The GLETQ measures number of bouts per week (0-7) of mild, moderate, or strenuous exercise that last at least 15 minutes.
Behavioral Risk Factor Surveillance System (BRFSS/2011) | Baseline
  Asks participants about meeting strength training guidelines (2 times per week)
Behavioral Risk Factor Surveillance System (BRFSS/2011) | 12 weeks
  Asks participants about meeting strength training guidelines (2 times per week)
Behavioral Risk Factor Surveillance System (BRFSS/2011) | 24 weeks
  Asks participants about meeting strength training guidelines (2 times per week)
Brief Pain Inventory (BPI) - Intensity and Interference | Baseline
  We will use the pain intensity and interference scales from the widely used BPI which uses a 0-10 Likert scale for ratings. A higher score indicates increased level of pain.
Brief Pain Inventory (BPI) - Intensity and Interference | 12 weeks
  We will use the pain intensity and interference scales from the widely used BPI which uses a 0-10 Likert scale for ratings. A higher score indicates increased level of pain.
Brief Pain Inventory (BPI) - Intensity and Interference | 24 weeks
  We will use the pain intensity and interference scales from the widely used BPI which uses a 0-10 Likert scale for ratings. A higher score indicates increased level of pain.
Positive (and Negative) Affect Schedule (PANAS) | Baseline
  The Positive (and Negative) Affect Schedule or (PANAS) is a scale that consists of 10 items with different words that describe feelings and emotion. - Adapted to use positive items only.
Positive (and Negative) Affect Schedule (PANAS) - Adapted to use positive items only | 12 weeks
  The Positive (and Negative) Affect Schedule or (PANAS) is a scale that consists of 10 items with different words that describe feelings and emotion. - Adapted to use positive items only.
Positive (and Negative) Affect Schedule (PANAS) - Adapted to use positive items only | 24 weeks
  The Positive (and Negative) Affect Schedule or (PANAS) is a scale that consists of 10 items with different words that describe feelings and emotion. - Adapted to use positive items only.
Patient Global Impression of Change (PGIC) | 12 weeks
  A 3-question scale designed to assess perception of change and improvement. The scale includes their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Patient Global Assessment of Treatment Satisfaction (PGATS) | 12 weeks
  A 1-question scale designed to assess satisfaction of treatment. It is scored from 0-10 or 0-100, with higher numbers representing worse perceived disease activity or overall health.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline
  The GAD-7 is a seven-item, self-report anxiety measure designed to assess health status during the previous 2 weeks. A higher score indicates a higher level of anxiety.
Generalized Anxiety Disorder-7 (GAD-7) | 12 weeks
  The GAD-7 is a seven-item, self-report anxiety measure designed to assess health status during the previous 2 weeks. A higher score indicates a higher level of anxiety.
Generalized Anxiety Disorder-7 (GAD-7) | 24 weeks
  The GAD-7 is a seven-item, self-report anxiety measure designed to assess health status during the previous 2 weeks. A higher score indicates a higher level of anxiety.
Quality of Life after Brain Injury Scale (QoLIBRI) | Baseline
  The QoLIBRI is a self-reported measure of satisfaction in areas including: thinking abilities, emotions, independence and social relationships and is a TBI Common Data Element measure. The QOLIBRI scores are reported on a 0-100 scale , where 0=worst possible quality of life and 100=best possible quality of life.
Quality of Life after Brain Injury Scale (QoLIBRI) | 12 weeks
  The QoLIBRI is a self-reported measure of satisfaction in areas including: thinking abilities, emotions, independence and social relationships and is a TBI Common Data Element measure. The QOLIBRI scores are reported on a 0-100 scale , where 0=worst possible quality of life and 100=best possible quality of life.
Quality of Life after Brain Injury Scale (QoLIBRI) | 24 weeks
  The QoLIBRI is a self-reported measure of satisfaction in areas including: thinking abilities, emotions, independence and social relationships and is a TBI Common Data Element measure. The QOLIBRI scores are reported on a 0-100 scale , where 0=worst possible quality of life and 100=best possible quality of life.
Patient Reported Outcomes Measurement Information System (PROMIS) 6 Item Fatigue Scale | Baseline
  The PROMIS 6a scale is composed of 6 items developed to assess the domain of sleep disturbances in the past 7 days.
Patient Reported Outcomes Measurement Information System (PROMIS) 6 Item Fatigue Scale | 12 weeks
  The PROMIS 6a scale is composed of 6 items developed to assess the domain of sleep disturbances in the past 7 days.
Patient Reported Outcomes Measurement Information System (PROMIS) 6 Item Fatigue Scale | 24 weeks
  The PROMIS 6a scale is composed of 6 items developed to assess the domain of sleep disturbances in the past 7 days.
Behavioral Activation for Depression Scale (BADS) | Baseline
  The BADS measure was developed to measure behavioral activation over the course of treatment. For all subscales, high scores are consistent with the subscale title.
Behavioral Activation for Depression Scale (BADS) | 12 weeks
  The BADS measure was developed to measure behavioral activation over the course of treatment. For all subscales, high scores are consistent with the subscale title.
Behavioral Activation for Depression Scale (BADS) | 24 weeks
  The BADS measure was developed to measure behavioral activation over the course of treatment. For all subscales, high scores are consistent with the subscale title.
Minutes per week of Moderate to Vigorous Physical Activity (MVPA) | Baseline
  We will use the Fitbit Charge 5 device settings and activity count cutoffs to measure moderate to vigorous physical activity (MVPA).
Minutes per week of Moderate to Vigorous Physical Activity (MVPA) | 12 weeks
  We will use the Fitbit Charge 5 device settings and activity count cutoffs to measure moderate to vigorous physical activity (MVPA).
Minutes per week of Moderate to Vigorous Physical Activity (MVPA) | 24 weeks
  We will use the Fitbit Charge 5 device settings and activity count cutoffs to measure moderate to vigorous physical activity (MVPA).

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bombardier, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the cycle prospectively collected study data for our module study will be completely de-identified and submitted to Inter-university Consortium for Political and Social Research (ICPSR). We intend to request that study data be embargoed for two years after the conclusion of the study(s) to allow enough time for study investigators to complete and disseminate the study aims. After that time, the data will be available publicly via ICPSR. The project will be assigned a DocID which will allow for persistent identification of the data and the project as a whole.
  chromeextension://efaidnbmnnnibpcajpcglclefindmkaj/https://acl.gov/sites/default/files/about-acl/2017-12/ACLPublicAcccessPlan.pdf
Supporting Information: Study Protocol, ICF
Time Frame: Scientific data will be made available to the public no later than 24 months after award end date of 08/31/2027.
Access Criteria: Administration of Community Living (ACL) (National Institute on Disability, Independent Living, and Rehabilitation Research (NIDILRR)) designates the Interuniversity Consortium for Political and Social Research (ICPSR), a unit within the Institute for Social Research at the University of Michigan that provides data archiving services, as its preferred data repository for scientific data from all ACL/NIDILRR-funded research. The exception to this designation is the archiving of longitudinal scientific data collected through the ACL/NIDILRR-funded Burn Injury, Spinal Cord Injury, and Traumatic Brain Injury Model Systems. For these three specific funding programs, the longitudinal scientific data have been and will continue to be deposited to and made publicly available by the National Statistical and Data Center of each respective model system. The National Statistical and Data Centers have the capacity to function as a data repository and making those data accessible to the public.
URL: https://www.icpsr.umich.edu/web/pages/datamanagement/confidentiality/conf-language.html

DOCUMENTS (1):
  • Informed Consent Form (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT06005194/ICF_000.pdf